CLINICAL TRIAL: NCT04835948
Title: Study of the Efficacy of Single Dose Anti-thymocyte Globulin in the Modulation of T Lymphocytes in Kidney Transplant Outcomes
Brief Title: Efficacy of Single Dose Anti-thymocyte Globulin in the Modulation of T Lymphocytes in Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabiani Palagi Machado, Principal Investigator, Hospital de Clinicas de Porto Alegre
Other Study IDs: 38361620.0.0000.5327
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Kidney Transplant; Complications; Immunosuppression
Keywords: Immunosuppression; kidney transplantation; CD3+ T lymphocytes; Anti-thymocyte globulin; Rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Antilymphocyte Serum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple doses of anti-thymocyte globulin (ATG): Control group that received fractionated doses of 1.5 mg/kg adding up to a total of 6 mg/kg
  Interventions: Drug: single dose of Anti-thymocyte globulin

INTERVENTIONS:
Drug: single dose of Anti-thymocyte globulin — Used anti-thymocyte globulin (ATG) in a single dose of 3 mg/kg for immunosuppression induction in the immediate postoperative period

SUMMARY:
The use of polyclonal anti-T cell antibodies (ATG) has benefits in kidney transplantation, however, its use is associated mainly with hematological, infectious, and neoplastic complications. Monitoring T cells in patients receiving ATG was first proposed in 1975 to improve efficacy in preventing acute rejection and avoiding excessive immunosuppression. The dose regimen is guided by a daily count of TCD3+ lymphocytes. Monitoring the dose of thymoglobulin through its biological effects on T cells is a rational and safe method of titrating the dose of that antibody. This way, it is possible to reduce the total amount of drug administered to the patient and, consequently, reduce undesirable complications, as well as the cost of treatment, without losing effect on the benefit of immunosuppression.

Currently, the usual cumulative dose of ATG for induction in kidney transplant patients is 6mg/kg, in divided doses. However, the ideal dose and duration of therapy are still the subject of studies, with protocols between centers varying from total doses of 3 to 6 mg/kg, either fractionated or single, to achieve the lowest dose with fewer undesirable effects, and with reduced length of inpatient stay.

The use of ATG in a single dose of 3 mg/kg was successfully assessed for risks of infection and rejection in patients with low immunological risk.

This study proposes evaluating the efficacy and safety of a single 3mg/kg dose of ATG for patients with low and standard immune risk, with TCD3+ lymphocyte monitoring, to assess the duration of the TCD3+ cells in the peripheral blood.

DETAILED DESCRIPTION:
Kidney transplantation is one of the major advances in medicine in the past 60 years. Currently, is considered the best treatment for terminal chronic kidney disease in the medium and long term, and the least costly. To obtain these successful outcomes, the immune response to the graft must be properly controlled and monitored since its implantation. T and B lymphocytes are crucial in the alloimmune response by mediating cellular and antibody-mediated rejections, respectively, and along with anti-HLA antibodies are the main effectors of acute and chronic rejections.

Anti-thymocyte globulin (ATG) has a key role in the immunosuppressive induction regimens used in kidney transplants as well as in the treatment of acute rejections. It is a purified solution that contains a variety of T cell-specific immunoglobulins, including CD2, CD3, CD4, CD8, CD11a, CD18, CD25, HLA-DR, and class I HLA (human leukocyte antigen). This solution is produced by immunizing rabbits with human thymocytes. The use of these agents is particularly important in inducing patients who are more predisposed to the nephrotoxic effects of calcineurin inhibitors (CI), allowing the delayed introduction of the CI. Induction with antibodies is also of great value in patients with higher immunological risk, such as pediatric, Afro-descendants, re-transplanted, and previously sensitized to HLA antigens recipients.

Polyclonal antibodies have definite benefits in kidney transplantation, but their use is associated with hematological, infectious, and neoplastic complications. The use of reduced doses of ATG has been the subject of recent studies, but still with inconclusive results.

The concept of monitoring T cells in patients receiving ATG was first proposed in 1975 to improve efficacy in preventing acute rejection and avoiding excessive immunosuppression. The dose regimen is guided by a daily count of peripheral blood TCD3+ lymphocytes. Monitoring the dose of thymoglobulin through its biological effects on T cells is a rational and safe method of titrating the dose of that antibody. This way, it is possible to reduce the total amount of drug administered to the patient and, consequently, reduce undesirable complications, as well as the cost of treatment, hopefully without losing effect on the benefit of immunosuppression.

A 60% reduction in the total dose of ATG and 58% reduction in therapy cost was observed in patients who were monitored using TCD3+ cell counts. Currently, the usual total dose of ATG for induction in kidney transplant patients is 6mg/kg, divided into 4 doses, which can be administered from day zero until day 14 (maximum) of transplantation. However, the ideal dose and duration of therapy are still the subject of investigation, with protocols between centers varying from total doses of 3 to 6 mg/kg, fractionated or single, to attempt to achieve the lowest dose with fewer undesirable effects, and with reduced length of inpatient stay. The use of ATG in a single dose of 3 mg/kg was successfully assessed for risks of infection and rejection in patients with low immunological risk.

Considering that the adverse effects associated with the use of ATG are relevant in the clinical context of kidney transplantation, the use of a lower dose, keeping its immunomodulatory effect, with a safer profile, is desirable.

The study evaluates the efficacy and safety of a single dose of 3mg/kg ATG for patients with low and standard immune risk, with TCD3+ lymphocyte monitoring, to assess the clinical efficacy and the modulation of the T cell response.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients from Hospital de Clínicas de Porto Alegre (HCPA) between October 2018 to March 2020 who received a single 3 mg/kg ATG dose at the immediate postoperative period. Recipients of standard and low immunological risk (PRA - panel reactive antibodies <50% and without donor-specific antibodies), regardless of the time of cold ischemia and the presence of kidney failure in the donor.
* Control group consisting of patients from the same and previous period, who received fractionated ATG dosing up to 6 mg/kg total dose.

Exclusion Criteria:

* Patients who used other induction strategies that did not include ATG in a single dose of 3 mg/kg or the fractionated dose of 6 mg/kg.
* Patients who died within 24 hours after transplantation.
* Patients who had a transplant nephrectomy within 24 hours after transplantation.
* Pediatric recipients (< 14 years old).
* Recipients with incomplete data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients who received a kidney transplant at a single institution between October 2018 and March 2020 and received ATG at a single dose of 3 mg/kg for induction of immunosuppression in the immediate postoperative period and a control group that received fractionated doses of 1.5 mg/kg adding up to a total of 6 mg/kg.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Immunomodulatory effect | one year
  Immunomodulatory effect of a single dose of 3mg/kg ATG on TCD3+ lymphocytes in kidney transplant patients by comparing it with the effect of the regular fractionated dose of 6 mg/kg by counting daily the number of TCD3+ lymphocytes in peripheral blood.

SECONDARY OUTCOMES:
Incidence of acute rejection | one year
  Number of patients with acute rejection diagnosed by renal biopsy with the single-dose ATG strategy.
Occurence of cytomegalovirus infection | One year
  Number of patients with cytomegalovirus infection (positive detection through polymerase chain reaction or active disease).
Incidence of delayed graft function | one year
  Number of patients with delayed graft function (DGF) through the number of dialysis needed in the first week after kidney transplantation.
One year survival of kidney grafts | One year
  Survival of kidney grafts at 1 year after receiving a single dose of ATG.
One year survival graft grafts | one year
  Patient survival at the end of 1 year of a single dose of ATG.

OTHER OUTCOMES:
Occurence of infections and neoplasms | One year
  Number of patients with development of other infections and neoplasms of any etiology within one year proven by clinical features and laboratory or anatomopathological tests in the study patients.
Hematological effects of the drug. | One year
  Number of patients with hematological effects (laboratory analysis of anemia, leukopenia and thrombocytopenia) of ATG.
Time of inpatient stay (days). | One year
  Length of stay in days between groups with a single and fractionated dose of atg.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nankivell BJ, Alexander SI. Rejection of the kidney allograft. N Engl J Med. 2010 Oct 7;363(15):1451-62. doi: 10.1056/NEJMra0902927. No abstract available. PMID 20925547
- [Background] Taylor DO, Kfoury AG, Pisani B, Hammond EH, Renlund DG. Antilymphocyte-antibody prophylaxis: review of the adult experience in heart transplantation. Transplant Proc. 1997 Dec;29(8A):13S-15S. doi: 10.1016/s0041-1345(97)00849-x. No abstract available. PMID 9414668
- [Background] First MR. Immunologically high-risk recipient strategies. Transplant Proc. 1999 Feb-Mar;31(1-2):243-6. doi: 10.1016/s0041-1345(98)01520-6. No abstract available. PMID 10083093
- [Background] Clesca P, Dirlando M, Park SI, Garcia R, Ferraz E, Pinheiro-Machado PG, Kushnaroff L, Tedesco-Silva H Jr, Medina-Pestana JO. Thymoglobulin and rate of infectious complications after transplantation. Transplant Proc. 2007 Mar;39(2):463-4. doi: 10.1016/j.transproceed.2007.01.024. PMID 17362760
- [Background] Gaber AO, Knight RJ, Patel S, Gaber LW. A review of the evidence for use of thymoglobulin induction in renal transplantation. Transplant Proc. 2010 Jun;42(5):1395-400. doi: 10.1016/j.transproceed.2010.04.019. PMID 20620442
- [Background] Djamali A, Turc-Baron C, Portales P, Leverson G, Chong G, Clot J, Mourad G. Low dose antithymocyte globulins in renal transplantation: daily versus intermittent administration based on T-cell monitoring. Transplantation. 2000 Mar 15;69(5):799-805. doi: 10.1097/00007890-200003150-00021. PMID 10755529
- [Background] Thiyagarajan UM, Ponnuswamy A, Bagul A. Thymoglobulin and its use in renal transplantation: a review. Am J Nephrol. 2013;37(6):586-601. doi: 10.1159/000351643. Epub 2013 Jun 12. PMID 23774740
- [Background] Alangaden GJ, Thyagarajan R, Gruber SA, Morawski K, Garnick J, El-Amm JM, West MS, Sillix DH, Chandrasekar PH, Haririan A. Infectious complications after kidney transplantation: current epidemiology and associated risk factors. Clin Transplant. 2006 Jul-Aug;20(4):401-9. doi: 10.1111/j.1399-0012.2006.00519.x. PMID 16842513
- [Background] Yang JW, Wang JN, Men TY, Zhang XM, Li XD, Shen B, Li GY, Chen DD. Comparison of clinical outcome of low-dose and high-dose rabbit antithymocyte globulin induction therapy in renal transplantation: a single-center experience. Ann Transplant. 2014 Jun 6;19:277-82. doi: 10.12659/AOT.890069. PMID 24906405
- [Background] Bishop G, Cosimi AB, Voynow NK, Whelchel JD, Wortis HH. Effect of immunosuppressive therapy for renal allografts on the number of circulating sheep red blood cells rosetting cells. Transplantation. 1975 Aug;20(2):123-9. doi: 10.1097/00007890-197508000-00005. PMID 1101478
- [Background] Wang CJ, Tuffaha A, Zhang D, Diederich DA, Wetmore JB. A CD3+ count-based thymoglobulin induction regimen permits delayed introduction of calcineurin inhibitors in kidney transplantation. Clin Transplant. 2012 Nov-Dec;26(6):900-9. doi: 10.1111/j.1399-0012.2012.01656.x. Epub 2012 Jun 4. PMID 22672562
- [Background] Peddi VR, Bryant M, Roy-Chaudhury P, Woodle ES, First MR. Safety, efficacy, and cost analysis of thymoglobulin induction therapy with intermittent dosing based on CD3+ lymphocyte counts in kidney and kidney-pancreas transplant recipients. Transplantation. 2002 May 15;73(9):1514-8. doi: 10.1097/00007890-200205150-00025. PMID 12023634
- [Background] Abouna GM, al-Abdullah IH, Kelly-Sullivan D, Kumar MS, Loose J, Phillips K, Yost S, Seirka D. Randomized clinical trial of antithymocyte globulin induction in renal transplantation comparing a fixed daily dose with dose adjustment according to T cell monitoring. Transplantation. 1995 Jun 15;59(11):1564-8. PMID 7778170
- [Background] Uber WE, Uber LA, VanBakel AB, Crumbley AJ 3rd, Pereira NL, Ikonomidis JS, Feldman DS. CD3 monitoring and thymoglobulin therapy in cardiac transplantation: clinical outcomes and pharmacoeconomic implications. Transplant Proc. 2004 Dec;36(10):3245-9. doi: 10.1016/j.transproceed.2004.11.099. PMID 15686739
- [Background] Krasinskas AM, Kreisel D, Acker MA, Bavaria JE, Pochettino A, Kotloff RM, Arcasoy S, Blumenthal N, Kamoun M, Moore JS, Rosengard BR. CD3 monitoring of antithymocyte globulin therapy in thoracic organ transplantation. Transplantation. 2002 Apr 27;73(8):1339-41. doi: 10.1097/00007890-200204270-00026. PMID 11981432
- [Background] Grandtnerova B, Mocikova H, Kohutova M. CD2+, CD3+, and CD19+ depletion after a course of antithymocyte globulin for a steroid-resistant rejection. Transplant Proc. 1997 Nov;29(7):2958-9. doi: 10.1016/s0041-1345(97)00744-6. No abstract available. PMID 9365628
- [Background] Kho MM, Bouvy AP, Cadogan M, Kraaijeveld R, Baan CC, Weimar W. The effect of low and ultra-low dosages Thymoglobulin on peripheral T, B and NK cells in kidney transplant recipients. Transpl Immunol. 2012 Jun;26(4):186-90. doi: 10.1016/j.trim.2012.02.003. Epub 2012 Mar 5. PMID 22410573
- [Background] Nafar M, Dalili N, Poor-Reza-Gholi F, Ahmadpoor P, Samadian F, Samavat S. The appropriate dose of thymoglobulin induction therapy in kidney transplantation. Clin Transplant. 2017 Jun;31(6). doi: 10.1111/ctr.12977. Epub 2017 Apr 18. PMID 28376289
- [Background] Tedesco-Silva H, Felipe C, Ferreira A, Cristelli M, Oliveira N, Sandes-Freitas T, Aguiar W, Campos E, Gerbase-DeLima M, Franco M, Medina-Pestana J. Reduced Incidence of Cytomegalovirus Infection in Kidney Transplant Recipients Receiving Everolimus and Reduced Tacrolimus Doses. Am J Transplant. 2015 Oct;15(10):2655-64. doi: 10.1111/ajt.13327. Epub 2015 May 18. PMID 25988935
- [Background] Mohty M, Bacigalupo A, Saliba F, Zuckermann A, Morelon E, Lebranchu Y. New directions for rabbit antithymocyte globulin (Thymoglobulin((R))) in solid organ transplants, stem cell transplants and autoimmunity. Drugs. 2014 Sep;74(14):1605-34. doi: 10.1007/s40265-014-0277-6. PMID 25164240
- [Background] Bauer AC, Franco RF, Manfro RC. Immunosuppression in Kidney Transplantation: State of the Art and Current Protocols. Curr Pharm Des. 2020;26(28):3440-3450. doi: 10.2174/1381612826666200521142448. PMID 32436821